CLINICAL TRIAL: NCT01472250
Title: A Prospective and Observational Cohort Study to Evaluate the Treatment Model and Medical Economics of Advanced Gastric Cancer Chemotherapy in Clinical Practice in China
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, chief of department of GI oncology, Peking University
Other Study IDs: CGOG1002
Record Dates: First submitted 2011-10-28; First posted 2011-11-16 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Advanced Gastric Cancer
Keywords: Advanced Gastric Cancer; chemotherapy; quality of life; treatment expense; patients accepted first-line chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the tumor tissue samples were collected to do gene mutation analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chemotherapy: Eligible patients will accept generalized chemotherapy according to the investigator's assessment.
  Interventions: Drug: Clinical chemo-drugs

INTERVENTIONS:
Drug: Clinical chemo-drugs — Clinical drugs will be selected by the investigator according to recommendations in Chinese and foreign guidelines and depending on clinical experience and the patient's individual conditions, including but not limited to the drugs listed below:
  Platinum products: oxaliplatin, cisplatin Fluorouracil products: 5-fluorouracil, capecitabine, TS-1 Taxanes: paclitaxel, docetaxel

SUMMARY:
This is a multi-center, prospective and observational clinical study. Eligible patients will accept generalized chemotherapy according to the investigator's assessment. Information related to the treatment, including medication, disease condition, expenses, etc. will be periodically collected. Follow-up at 2-month intervals will be periodically performed to continually collect information about the disease progression, subsequent treatment and survival until death or completion of the study.

Recruited patients will fill out questionnaires about quality of life before initiation of treatment, at Cycle 3 and completion of first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has histologically confirmed locally-advanced or recurrent and/or metastatic gastric or esophagogastric junction adenocarcinoma, has missed the opportunity of surgical excision, making curative therapy impossible.
2. The informed consent form is signed.
3. A specimen of tumor tissue (puncture biopsy or surgical specimen) is available.
4. ECOG performance status is 0, 1 or 2.
5. The patient's general conditions and functions of important organs allow generalized chemotherapy according to the investigator's judgment
6. The patient is aged≥18

Exclusion Criteria:

1. The patient is known to be allergic to any study drug.
2. The patient is recruited in other clinical study or is planned to participate into other clinical study.
3. The patient has previously accepted chemotherapy against advanced or metastatic diseases (the patient may be recruited if the previous adjuvant therapy/neoadjuvant therapy was completed more than 6 months before inclusion).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2011-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
chemotherapy regimen | 2 months
  To evaluate the treatment model (singel or doublet or triplet chemotherapy)of patients with advanced gastric cancer in China

SECONDARY OUTCOMES:
overall survival | 2 months
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 2 months till death or lost
quality of life | 6 weeks
  To evaluate the quality of life before and after chemotherapy of Chinese patients in real clinical practice
treatment expense | 2 months
  To evaluate the treatment expense of first-line treatment of Chinese patients with advanced gastric cancer in real clinical practice

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Shen, Beijing, Beijing Municipality, China